CLINICAL TRIAL: NCT00679185
Title: Effects of Expressive Writing in Breast Cancer Survivors With Lymphedema
Brief Title: Expressive Writing in Improving Quality of Life in Patients With Breast Cancer and Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sheila Ridner, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000587736; VU-VICC-SUPP-0422; NCT00400049 (obsolete NCT alias)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Fatigue; Lymphedema
Keywords: fatigue; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental-EW (Experimental): four emotion focused writing assignments
  Interventions: Behavioral: expressive writing
- control group (Active Comparator): non-emotional writing control
  Interventions: Behavioral: expressive writing

INTERVENTIONS:
Behavioral: expressive writing — four non-emotional writing assignments
  Other Names: none noted

SUMMARY:
RATIONALE: Expressive writing may help relieve symptoms and improve quality of life in breast cancer survivors with chronic lymphedema.

PURPOSE: This clinical trial is studying expressive writing in improving the quality of life in women with breast cancer and lymphedema.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if expressive writing improves quality of life (QOL) relative to the control condition in breast cancer survivors with chronic stage II lymphedema.
* To determine if expressive writing improves physical and psychological symptoms/outcomes (i.e., fatigue, psychological distress, activity level, confidence in body) relative to the control condition in breast cancer survivors with chronic lymphedema.

Secondary

* To explore the influence of individual difference variables (dispositional optimism, emotional intelligence, and repressive coping) on outcomes associated with this intervention to include identification of subsets of individuals for whom expressive writing is most effective.
* To explore the influence of intrusive/avoidant thinking as a mediator between the intervention and outcomes of QOL and physical and psychological symptoms.

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

Patients travel to the School of Nursing at Vanderbilt University or meet a team member in their home or another private location for an initial visit. Patients complete questionnaires, are measured for height and weight data, and arm fluid measurements.

* Expressive writing group: Twenty minutes a day, twice a week for 2 weeks, patients write about their deepest thoughts and feelings regarding their lymphedema and its treatment.
* Daily diary group (control): Twenty minutes a day, twice a week for 2 weeks patients write about how they manage their time .

Patients complete quality-of-life questionnaires periodically.

After completion of study, patients are followed at 1, 3, and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women who have undergone prior surgery and/or radiotherapy for breast cancer

  * No metastatic disease
* Must have lymphedema, meeting the following conditions:

  * Stage II disease

    * Swelling unrelieved by elevation, arm may be hard, may not pit with pressure, or skin changes have taken place
  * Received prior professional treatment for lymphedema
  * Requires life-long, at home self-care (e.g., compression sleeves)
* No history of bilateral lymphedema prohibiting extracellular fluid comparison to an unaffected limb

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Able to read, write (for 20 minutes), and speak English
* Willing and able to drive to the study site or agree to be seen in an outpatient setting (e.g., private therapist office, outpatient clinic, physicians office, or own home) once

Exclusion criteria:

* Has medical condition that could cause edema, including any of the following:

  * Symptomatic congestive heart failure
  * Chronic/acute renal disease
  * Cor pulmonale
  * Nephrotic syndrome
  * Nephrosis
  * Liver failure
  * Cirrhosis
  * Pregnant or expect to become pregnant during course of the study
* Unable to stand upright for measurement of height and weight
* Has a metal implant, internal defibrillator, or pacemakers
* History of suicide attempts
* No recent suicidal ideation (within last 6 months)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent intravenous chemotherapy or radiotherapy for active cancer
* No concurrent antipsychotic medication (i.e., haldol, thorazine, stelazine)

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Physical and psychological symptoms | 6 months
Quality of life | 6 months
Fatigue | 6 months
Psychological distress | 6 months
Activity level | 6 months

SECONDARY OUTCOMES:
Influence of intrusive/avoidant thinking in quality of life and physical or psychological symptoms | baseline study entry
Influence of individual difference variables to discover subsets for treatment effectiveness | baseline study entry

CONTACTS AND LOCATIONS:
Overall Officials: Shiela H. Ridner, MSHSA, MSN, PhD, RN, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Ridner SH, Bonner CM, Deng J, Sinclair VG. Voices from the shadows: living with lymphedema. Cancer Nurs. 2012 Jan-Feb;35(1):E18-26. doi: 10.1097/NCC.0b013e31821404c0. PMID 21558848